CLINICAL TRIAL: NCT01827969
Title: Feasibility Study of Ablathermy Focused Ultrasound (USF) of Breast Tumors Before Mastectomy
Acronym: USF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IB2009-58
Record Dates: First submitted 2012-11-06; First posted 2013-04-10 (Estimated); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Breast Tumor
Keywords: Women; breast tumor; planned mastectomy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ablathermy focused ultrasound (Experimental): ablathermy focused ultrasound
  Interventions: Procedure: ablathermy focused ultrasound

INTERVENTIONS:
Procedure: ablathermy focused ultrasound — ablathermy focused ultrasound

SUMMARY:
The treatment consists of tumor ablation by Ablathermy Focused Ultrasound (USF), guided by MRI, performed under local anesthesia and sedation.

DETAILED DESCRIPTION:
The treatment consists of tumor ablation by USF, guided by MRI, performed under local anesthesia and sedation. Patients will be operated (mastectomy) from 48 hours after ablation.

ELIGIBILITY:
Inclusion Criteria:

* Invasive Breast Carcinoma with histologically confirmed hormone receptor analysis, the grade of the tumor, the expression of Her-2.
* Lesion classified T1-T2-T3 unifocal or multifocal with or without associated microcalcifications
* Lesion recognizable and identifiable in MRI
* Indication of mastectomy with or without axillary
* Lesion located more than 10 mm from the skin, the nipple and pectoralis major
* No cons-indication to MRI (pacemaker)
* Women whose age is ≥ 18 years
* If premenopausal patient: patient contraceptives
* Patient has signed informed consent
* Affiliation to a social security scheme

Exclusion Criteria:

* Tumor-TD T4B classified or non-palpable lesion
* If age <70 years: no indication of adjuvant chemotherapy and neoadjuvant
* MRI lesions have not been identified, located within 10 mm of the skin and pectoral muscle, greater than 25 mm diameter
* Inability to hold still in the prone position, arms extended, for 30 minutes
* Contraindication to MRI
* Patient deprived of liberty and major subject of a measure of legal protection or unable to consent
* Patient participating in another interventional clinical trial within 30 days prior to baseline and during the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Effectiveness of ablathermy | 2 years
  Effectiveness of ablathermy focused ultrasound breast tumors will be assessed based on histological criteria : the intervention will be considered effective for a participant if there is a destruction of the tumor mass by coagulation necrosis

CONTACTS AND LOCATIONS:
Overall Officials: PALUSSIERE Jean, MD, Study Chair — Institut Bergonié
Locations (1):
- Institut Bergonié, Bordeaux, Aquitaine, France

IPD SHARING:
Plan to Share IPD: No